CLINICAL TRIAL: NCT00768248
Title: Ambulatory Continuous Peripheral Nerve Blocks for Treatment of Post-Amputation Phantom Limb and Stump Pain
Brief Title: Naval Medical Center San Diego (NMCSD) - Ambulatory Continuous Peripheral Nerve Blocks for Treatment of Post-Amputation Phantom Limb and Stump Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No longer enrolling patients, not enough enrollment
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Associate Professor, In Residence, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NMCSD Phantom Pilot
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Results first posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-07

CONDITIONS: Amputation; Phantom Limb; Stump Pain
Keywords: pain; phantom limb; stump pain; catheter; nerve block; peripheral nerve block; NMCSD; Post-Amputation Phantom Limb or Stump Pain
MeSH Terms: conditions — Phantom Limb; Pain | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Active Comparator): 3-7 days of perineural local anesthetic infusion
  Interventions: Drug: perineural ropivacaine
- Placebo (Placebo Comparator): 3-7 days of perineural normal saline infusion
  Interventions: Drug: normal saline (placebo)

INTERVENTIONS:
Drug: perineural ropivacaine — ropivacaine 0.4%; the basal rate will be set at 7 mL/h
  Arms: Active
Drug: normal saline (placebo) — the basal rate will be set at 7 mL/h
  Arms: Placebo

SUMMARY:
The purpose of this research study is to determine if putting local anesthetic-or numbing medication-through one or two tiny tube(s) placed next to the nerves that go to an amputated limb will decrease phantom limb and/or stump pain.

DETAILED DESCRIPTION:
Specific Aim 1: To determine if, compared with current standard-of-care treatment, the addition of an ambulatory continuous peripheral nerve block decreases post-amputation phantom limb and stump pain.

Hypothesis 1: Following upper or lower extremity amputation, phantom limb and/or stump pain will be significantly decreased four weeks following a multiple-day ambulatory continuous peripheral nerve block as compared with patients receiving standard-of-care treatment (as measured on the 11-point numeric rating scale).

Specific Aim 2: To investigate the possible relationship between the addition of a multiple-day ambulatory continuous peripheral nerve block to standard-of-care treatment of post-amputation phantom limb and/or stump pain and cortical reorganization.

Hypothesis 2: Following upper or lower extremity amputation with subsequent phantom limb pain/sensation and/or stump pain, the addition of a multiple-day ambulatory continuous peripheral nerve block to standard-of-care treatment will result in cortical reorganization during and four-weeks following the perineural infusion (as measured by MRI).

ELIGIBILITY:
Inclusion Criteria:

* previous upper or lower limb amputation including at least one metacarpal or metatarsal bone, respectively
* age 18 years or older
* phantom limb and/or stump pain described as at least a 2 on the NRS for the previous week [and pain occurring on a weekly basis over the previous month]
* willing to have an ambulatory perineural infusion for 6 days
* willing to avoid additional "new" analgesic interventions from 4 weeks prior to at least 4 weeks following catheter placement, and preferably to 6 months following catheter placement
* the availability of a "caretaker" who will transport the subject home following the procedure and remain with the subject for the first night of the infusion

Exclusion Criteria:

* known hepatic or renal insufficiency
* allergy to the study medications
* possessing a contraindication to perineural catheter placement or perineural local anesthetic infusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Hanling, M.D., Principal Investigator — United States Naval Medical Center, San Diego
Locations (1):
- Naval Medical Center San Diego, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment failed at this center (NMCSD)--two subject were enrolled but they did not have data collected [coordinator simply did not collect the data] and so this pilot study was closed without producing results.
Period: Overall Study
Arm/Group | Active | Placebo
Started | 1 | 1
Completed | 0 | 0
Not Completed | 1 | 1
Not completed — Research coordinator didn't collect data | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Placebo | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 24 [24 to 24] | 23 [23 to 23] | 23.5 [23.5 to 23.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Primary Analysis Will Compare the Two Treatment Groups for the Phantom Limb/Stump Pain Change From Baseline to 4 Weeks Following the Initial Catheter Placement
Time Frame: Week 4
Population: Recruitment failed at this center (NMCSD)--two subject were enrolled but they did not have data collected [coordinator simply did not collect the data] and so this pilot study was closed without producing results.
Arm/Group | Active | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Physical Functioning · Brief Pain Inventory
Time Frame: pre-intervention, then days 1, 3, 8, 28, 84, and 365
Population: as for outcome 1
Arm/Group | Active | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Emotional Functioning · Beck Depression Inventory
Time Frame: pre-intervention; and then day 28 and 365 post-intervention
Population: as for outcome 1
Arm/Group | Active | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Nervous System Reorganization [if Patient Elected to Participate in the MRI Procedures] · MRI Procedure
Time Frame: pre-intervention; and then 8 and 28 days post-intervention
Population: as for outcome 1
Arm/Group | Active | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Pain · 11-point Numeric Rating Scale of Pain Intensity · Usage of Baseline and Rescue Analgesics in Previous 24 Hours · Patient Global Impression of Change Scale
Time Frame: Day 8, Day 28, Month 12
Population: as for outcome 1
Arm/Group | Active | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: not collected: Recruitment failed at this center (NMCSD)--two subject were enrolled but they did not have data collected [coordinator simply did not collect the data] and so this pilot study was closed without producing results.
Description: Recruitment failed at this center (NMCSD)--two subject were enrolled but they did not have data collected [coordinator simply did not collect the data] and so this pilot study was closed without producing results.
Arm/Group | Active | Placebo
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes